CLINICAL TRIAL: NCT02825199
Title: Effect of Caffeine Intake in Vestibular Function: A Randomized Triple-Blind Controlled Trial
Brief Title: Effect of Caffeine Intake in Vestibular Function
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto Brasiliense de Otorrinolaringologia (Other)
Responsible Party: Principal Investigator, Alleluia Lima Losno Ledesma, Audiologist, Instituto Brasiliense de Otorrinolaringologia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: IBOtorrinolaringologia
Record Dates: First submitted 2016-06-08; First posted 2016-07-07 (Estimated); Last update posted 2016-07-07 (Estimated); Status verified 2016-07

CONDITIONS: Vertigo; Diseases, Vestibular; Caffeine
MeSH Terms: conditions — Vertigo; Vestibular Diseases | interventions — Caffeine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Caffeine group (Experimental): All participants underwent otoscopy and tympanometry, responded to the Profile of Mood State (POMS), submitted to the cVEMP, oVEMP and caloric tests in that order. After that they received caffeine capsule (300mg). After 45 minutes they again responded to the POMS, repeated the cVEMP, oVEMP and caloric test.
  Interventions: Dietary Supplement: Caffeine
- Non caffeine group (Placebo Comparator): All participants underwent otoscopy and tympanometry, responded to the Profile of Mood State (POMS), submitted to the cVEMP, oVEMP and caloric tests in that order. After that they received placebo capsule (maize starch). After 45 minutes they again responded to the POMS, repeated the cVEMP, oVEMP and caloric test.
  Interventions: Dietary Supplement: Non caffeine

INTERVENTIONS:
Dietary Supplement: Caffeine — capsule: 300mg caffeine
  Arms: Caffeine group
Dietary Supplement: Non caffeine — capsule: placebo (maize starch)
  Arms: Non caffeine group

SUMMARY:
Objective: Assess the effect of caffeine in the following vestibular function tests: Cervical Vestibular Evoked Potential (cVEMP), Ocular Vestibular Evoked Potential(oVEMP) and Caloric Test.

Methods: Randomized, prospective triple-blind, placebo controlled clinical trial. All participants underwent otoscopy, tympanometry, responded to the Profile of Mood State (POMS), submitted to the cVEMP, oVEMP and caloric tests. After that they received placebo or caffeine capsule (300mg) and repeated the procedures 45 minutes after.

DETAILED DESCRIPTION:
Trial design

This is a randomized, prospective triple-blind, placebo controlled clinical trial approved by the institutional review board under protocol number 1.399.322/16. Informed consent was obtained after a full explanation of the experimental procedure.

Participants

The sample was made up of medical students who agreed to participate as volunteers and had no hearing and/or vestibular complaints or other health problems that could affect the homeostasis of the vestibular system (problems in the cervical spine, cardiovascular problems, migraine, metabolic disorders, hormonal changes, psychiatric disorders, neurological diseases, use of prescription drugs continuously, smokers, alcoholics, illegal drug users).

Randomization, allocation and Blinding

At baseline, study participants were randomized to receive caffeine or placebo at a 1:1 ratio, by independent statistician. Was used a completely randomized design for two treatments which PLAN procedure (SAS 9.4). The allocation was made for a person outside the study what identified the capsules in identical packages labeled with the name of the participants. The active (caffeine) and placebo (maize starch) capsules were identical in color, size, weight, and packaging.

Interventions

All participants underwent otoscopy and tympanometry, responded to the Profile of Mood State (POMS), submitted to the cVEMP, oVEMP and caloric tests in that order. After that the participants received placebo or caffeine capsule (300mg). After 45 minutes the subjects again responded to the POMS, repeated the cVEMP, oVEMP and caloric test. The tests were performed in a center of rehabilitation of hearing and balance for the same audiologist, with the data collection period was 3 months.

Caffeine consumption

To determine caffeine consumption a questionnaire which sought to investigate eating habits was applied. The participants have to include for each item (coffee, teas, soft drinks, chocolate, powdered chocolate, powdered guarana, food supplements and energy drink) the amount, kind (i.e. espresso, filter coffee) and brand. Based on these data, the consumption was calculated using a preview standardization. From there, the subjects were classified according to consumption: sporadic (less than 100mg), light (100 to 299mg), moderate (300 to 499mg). Those who had higher intakes equal to 500mg / day or more (heavy or very heavy) were excluded.

POMS

Self-administered instrument that consists of 65 items describing feelings; to them should be assigned values from 0 to 4 according to the Likert scale of 5 points (0 -no, 1 - a little, 2 - more or less, 3 - well, 4 - extremely). The POMS aims to evaluate six factors: tension-anxiety (9 items), depression-dejection (15 items), anger-hostility (12 items), vigor-activity (8 items), fatigue-inertia (7 items), confusion-bewilderment (7 items), and a total mood disturbance score (TMD)

cVEMP

VEMP was performed in response to air-conducted stimuli, using alternate 500Hz (Hertz) tone bursts presented at 120 dB (decibel) and rate of 5.1 stimuli per second. Bandpass filter of 10 Hz to 1500 Hz was used, 50ms window and 200 stimulations in each track were standard. Two stimulations were recorded on each side, in order to observe the replicability. The stimuli were presented via insert earphones. A cleaning of the skin with abrasive paste was performed and surface electrodes were affixed using conductive paste. The non inverting electrode was placed in the middle part of the sternocleidomastoid, the ground electrode in lower forehead and the inverting on the upper forehead. The impedance of the electrodes should be less than or equal to 5hms. Subjects were positioned seated and instructed to maintain maximum head turn to the side contralateral to the stimulus throughout stimulation.The latency of P1 and N1 and the P1N1 amplitude were analyzed in each ear and an asymmetry rate was also analyzed. For the last one was used the formula: ǀ amplitude of right ear ǀ - ǀ amplitude of left ear ǀ / ǀ amplitude of right ear ǀ + ǀ amplitude of left ear ǀ x 100. To compare the amplitudes in each ear before and after tests was used the rate of change formula, consisting of: ǀ amplitude of ear before ǀ - ǀ amplitude of ear after ǀ / ǀ amplitude of ear before ǀ + ǀ amplitude of ear after ǀ x 100. The investigators considered normal p13 latencies between 13.9 to 19.2 and from 22.9 to 30.3 n23 and the asymmetry rate and rate of change of up to 28%.

oVEMP

The investigators used the same parameters of stimulation and analysis described in cVEMP. Non inverting electrodes were placed on the face just inferior to each eye (inferior oblique muscle), reference electrode was placed 1-2cm below contralateral to the stimulus and ground electrode in the forehead. The subject was placed in the sitting position and instructed to look upward. The latencies of initial negative (nI) and positive (pI) peak were measured. They considered normal nI latencies from 10.2 to 11.8 and from 14.7 to17.3 pI.

Caloric test

To perform the caloric test the investigators used an air otocalorimeter, and carried out four stimulations of 60 seconds each, with a flow of 8 liters per minute: 50C in the right ear, 50C on the left, 24C on the left ear and 24C in the right ear, in this order. The absolute values and percentages of unilateral weakness or directional preponderance were analyzed for each subject in each test. The subjects were considered normal when they showed absolute values from 3 to 45, a range of 30% or less in directional preponderance and of less than 25% in the unilateral weakness.

Outcomes

The primary outcome was the latency waves for cVEMP and oVEMP and absolute and relative values for caloric tests. These parameters were chosen for analysis of the primary outcome for being these the most well-established parameters for use in clinical practice. The secondary outcomes were asymmetry ratio and ratio of change for cVEMP. There were no secondary outcomes for oVEMP and Caloric test.

Statistical analysis

Non-parametric tests were used seeking statistically describe and compare the two groups - caffeine and no caffeine (Mann-Whitney test), the two time points - before and after in each group (Wilcoxon signed-rank test) and study the statistical effect of caffeine consumption on the other variables (Jonckheere-Terpstra test). It was used a confidence interval of 95%.The spreadsheet MS-Excel was used in your version of MS-Office 2013, for the organization of data, and IBM SPSS (International Business Machines - Statistical Package for Social Sciences), in its version 23.0, to obtain the results.

ELIGIBILITY:
Inclusion Criteria:

* Medical students volunteers
* Had no hearing and/or vestibular complaints

Exclusion Criteria:

* Problems in the cervical spine
* Cardiovascular problems
* Migraine
* Metabolic disorders
* Hormonal changes
* Psychiatric disorders
* Neurological diseases
* Use of prescription drugs continuously
* Smokers
* Alcoholics
* Illegal drug users

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2016-02; Primary Completion 2016-04 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
wave latency - VEMP | through study completion, an average of 3 months
asymmetry rate - VEMP | through study completion, an average of 3 months
Peak slow velocity (PSV) - Caloric test | through study completion, an average of 3 months
Unilateral weakness or directional preponderance - Caloric test | through study completion, an average of 3 months

SECONDARY OUTCOMES:
Questionnaire - POMS | through study completion, an average of 3 months
  Total of Mood Sates - It is a numerical scale that describes the participant's mood at that moment

CONTACTS AND LOCATIONS:
Overall Officials: Alleluia Ledesma, Audiologist, Principal Investigator — Instituto Brasiliense de Otorrinolaringologia
Locations (1):
- Instituto Brasiliense de Otorrinolaringologia (IBORL), Brasília, Federal District, Brazil

IPD SHARING:
Plan to Share IPD: Yes
The data will be published in full on the master's dissertation

REFERENCES:
- [Background] Akin FW, Murnane OD, Proffitt TM. The effects of click and tone-burst stimulus parameters on the vestibular evoked myogenic potential (VEMP). J Am Acad Audiol. 2003 Nov;14(9):500-9; quiz 534-5. doi: 10.3766/jaaa.14.9.5. PMID 14708838
- [Background] Akin FW, Murnane OD, Panus PC, Caruthers SK, Wilkinson AE, Proffitt TM. The influence of voluntary tonic EMG level on the vestibular-evoked myogenic potential. J Rehabil Res Dev. 2004 May;41(3B):473-80. doi: 10.1682/jrrd.2003.04.0060. PMID 15543465
- [Background] Felipe L, Santos MA, Goncalves DU. Vestibular evoked myogenic potential (Vemp): evaluation of responses in normal subjects. Pro Fono. 2008 Oct-Dec;20(4):249-54. doi: 10.1590/s0104-56872008000400008. PMID 19142468
- [Background] Carnauba AT, Lins OG, Soares Ido A, Andrade KC, Menezes Pde L. The impact of stimulation rates in vestibular evoked myogenic potential testing. Braz J Otorhinolaryngol. 2013 Sep-Oct;79(5):594-8. doi: 10.5935/1808-8694.20130106. PMID 24141674
- [Background] Lim CL, Clouston P, Sheean G, Yiannikas C. The influence of voluntary EMG activity and click intensity on the vestibular click evoked myogenic potential. Muscle Nerve. 1995 Oct;18(10):1210-3. doi: 10.1002/mus.880181021. No abstract available. PMID 7659119
- [Background] Wu CH, Young YH, Murofushi T. Tone burst-evoked myogenic potentials in human neck flexor and extensor. Acta Otolaryngol. 1999;119(7):741-4. doi: 10.1080/00016489950180351. PMID 10687928
- [Background] Welgampola MS, Colebatch JG. Characteristics and clinical applications of vestibular-evoked myogenic potentials. Neurology. 2005 May 24;64(10):1682-8. doi: 10.1212/01.WNL.0000161876.20552.AA. PMID 15911791
- [Background] Blakley BW, Wong V. Normal Values for Cervical Vestibular-Evoked Myogenic Potentials. Otol Neurotol. 2015 Jul;36(6):1069-73. doi: 10.1097/MAO.0000000000000752. PMID 25839981
- [Background] Rosengren SM, Govender S, Colebatch JG. Ocular and cervical vestibular evoked myogenic potentials produced by air- and bone-conducted stimuli: comparative properties and effects of age. Clin Neurophysiol. 2011 Nov;122(11):2282-9. doi: 10.1016/j.clinph.2011.04.001. Epub 2011 May 6. PMID 21550301
- [Background] Chihara Y, Iwasaki S, Ushio M, Murofushi T. Vestibular-evoked extraocular potentials by air-conducted sound: another clinical test for vestibular function. Clin Neurophysiol. 2007 Dec;118(12):2745-51. doi: 10.1016/j.clinph.2007.08.005. Epub 2007 Oct 1. PMID 17905655